CLINICAL TRIAL: NCT00018889
Title: Phenotype/Genotype Correlations in Movement Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010206; 01-N-0206
Record Dates: First submitted 2001-07-07; First posted 2001-07-09 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-11-07

CONDITIONS: Movement Disorder
Keywords: Clinical Evaluation; Genetic Study; Essential Tremor; Familial Myoclonus; Hereditary Ataxia; Natural History; Movement Disorder; Inherited Movement Disorder
MeSH Terms: conditions — Movement Disorders; Essential Tremor; Spinocerebellar Degenerations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients 1: Patients with diseases of known molecular basis will be genotyped in order to investigate phenotype/genotype correlations.
- Patients 2: Patients with disease of unknown or incomplete genetic characterization.
- Subjects: Subjects older than 2 years old with movement disorders and their family members

SUMMARY:
The goal of this protocol is to identify families with inherited movement disorders and evaluate disease manifestations to establish an accurate clinical diagnosis by using newest technological advances and investigate the underlying molecular mechanisms. Studies of inherited movement disorders in large families with good genealogical records are especially valuable. Patients with diseases of known molecular basis will be genotyped in order to investigate phenotype/genotype correlation. Patients with disease of unknown or incomplete genetic characterization will be studied with a hope of contributing to the identification of specific disease-causing genes and genetic mechanisms responsible for a specific disorder.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to perform phenotypic and genotypic characterizations of patients and family members with a known or suspected diagnosis of a movement disorder and screen for eligibility to participate in other movement disorder related protocols:

* 14-N-0086 Deep brain stimulation therapy in movement disorders
* 11-N-0211 Deep brain stimulation surgery for movement disorders
* 000865: Natural history of movement disorders
* 00-N-0043: Clinical and molecular manifestations of inherited neurologic disorders
* 03-AG-N-329 (NIA): The genetic characterization of movement disorders and dementias
* 20M0082 Phase 1 Study: PET Imaging of Cyclooxygenases in Neurodegenerative Brain Disease; Institute (NIMH)

The secondary goals of this protocol are to learn more about genetic causes of movement disorders and their phenotypic associations; identify patients and families with inherited movement disorders; evaluate disease manifestations to establish an accurate clinical diagnosis; and to investigate the underlying molecular mechanisms. Studies of inherited movement disorders in large families with well-documented genealogical records are especially valuable. The study will also assess a series of exploratory peripheral biomarkers, including, but not limited to, those delineated by DNA, RNA, protein, and/or metabolite alterations in an effort to more accurately predict those with, or at risk of having, the specific neurological disease.

Study population: Subjects older than 2 years old with movement disorders and their family members will be enrolled. Patients with diseases of known molecular basis will be genotyped in order to investigate phenotype/genotype correlations. Patients with disease of unknown or incomplete genetic characterization will be studied with a hope of contributing to the identification of specific disease-causing genes and genetic mechanisms and/or peripheral bio-signatures involved in a particular disorder.

Design:

This is an observational diagnostic study of movement disorders and their progression and pathophysiology.

Outcome measures: Determination of phenotype/genotype correlations in specific movement disorders, referral of patients and/or family members for participation in other NIH studies, gene identification if not known, gene expression and protein, metabolite and nucleic acid levels, collection of blood cells and generation of induced pluripotent stem cell lines, and establishment of a clinical diagnosis when possible.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals with suspected movement disorders
* Family members of movement disorders patients
* Ability to give informed consent or have a legally authorized representative able to give consent (for adults without consent capacity) or parent/guardian able to provide informed consent (for a child)
* If unable to give informed consent, ability to give assent (for children or adults without consent capacity)
* NIH Employees can participate in this study if they meet eligibility.

EXCLUSION CRITERIA:

* Pregnant women
* Children less than 2 years of age
* Employees of the Parkinson's Disease Clinic, NINDS

Exclusion criteria for MRI

* Presence of metal in subject s body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if subject was a welder or metal worker, since small metal fragments in the eye may be present.
* Subject is uncomfortable in small closed spaces (have claustrophobia) so that they would feel uncomfortable in the MRI machine.
* Unable to lie comfortably on back for up to 1 hour
* Under 12 years of age

There is no general exclusion for NIH employees.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects older than 2 years old with movement disorders and their family members will be enrolled. Patients with diseases of known molecular basis will be genotyped in order to investigate phenotype/genotype correlations. Patients with disease of unknown or incomplete genetic characterization will be studied with a hope of contributing to the identification of specific disease-causing genes and genetic mechanisms and/or peripheral bio-signatures involved in a particular disorder.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2001-10-22 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the phenotypic and genotypic characterizations of patients and family members with movement disorders. | 10 Years
  Characterizations to determine their eligibility for inclusion in other NIH protocols.

SECONDARY OUTCOMES:
Identification of disease-specific biomarkers in stem cells derived from patient peripheral blood mononuclear cells or fibroblast lines | Study end
Identification of new genes and/or peripheral blood biomarkers associated with movement disorders | Study end
Identification of new genes and/or peripheral blood biomarkers associated with movement disorders. | Study end
Establishment of a clinical diagnosis (when possible) | Study end
Referral of patients and/or family members for participation in other NIH studies | Study end

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Since this protocol is primarily a screening protocol, it may not be feasible to make data available on an individual patient level.

REFERENCES:
- [Background] Venter JC, Adams MD, Myers EW, Li PW, Mural RJ, Sutton GG, Smith HO, Yandell M, Evans CA, Holt RA, Gocayne JD, Amanatides P, Ballew RM, Huson DH, Wortman JR, Zhang Q, Kodira CD, Zheng XH, Chen L, Skupski M, Subramanian G, Thomas PD, Zhang J, Gabor Miklos GL, Nelson C, Broder S, Clark AG, Nadeau J, McKusick VA, Zinder N, Levine AJ, Roberts RJ, Simon M, Slayman C, Hunkapiller M, Bolanos R, Delcher A, Dew I, Fasulo D, Flanigan M, Florea L, Halpern A, Hannenhalli S, Kravitz S, Levy S, Mobarry C, Reinert K, Remington K, Abu-Threideh J, Beasley E, Biddick K, Bonazzi V, Brandon R, Cargill M, Chandramouliswaran I, Charlab R, Chaturvedi K, Deng Z, Di Francesco V, Dunn P, Eilbeck K, Evangelista C, Gabrielian AE, Gan W, Ge W, Gong F, Gu Z, Guan P, Heiman TJ, Higgins ME, Ji RR, Ke Z, Ketchum KA, Lai Z, Lei Y, Li Z, Li J, Liang Y, Lin X, Lu F, Merkulov GV, Milshina N, Moore HM, Naik AK, Narayan VA, Neelam B, Nusskern D, Rusch DB, Salzberg S, Shao W, Shue B, Sun J, Wang Z, Wang A, Wang X, Wang J, Wei M, Wides R, Xiao C, Yan C, Yao A, Ye J, Zhan M, Zhang W, Zhang H, Zhao Q, Zheng L, Zhong F, Zhong W, Zhu S, Zhao S, Gilbert D, Baumhueter S, Spier G, Carter C, Cravchik A, Woodage T, Ali F, An H, Awe A, Baldwin D, Baden H, Barnstead M, Barrow I, Beeson K, Busam D, Carver A, Center A, Cheng ML, Curry L, Danaher S, Davenport L, Desilets R, Dietz S, Dodson K, Doup L, Ferriera S, Garg N, Gluecksmann A, Hart B, Haynes J, Haynes C, Heiner C, Hladun S, Hostin D, Houck J, Howland T, Ibegwam C, Johnson J, Kalush F, Kline L, Koduru S, Love A, Mann F, May D, McCawley S, McIntosh T, McMullen I, Moy M, Moy L, Murphy B, Nelson K, Pfannkoch C, Pratts E, Puri V, Qureshi H, Reardon M, Rodriguez R, Rogers YH, Romblad D, Ruhfel B, Scott R, Sitter C, Smallwood M, Stewart E, Strong R, Suh E, Thomas R, Tint NN, Tse S, Vech C, Wang G, Wetter J, Williams S, Williams M, Windsor S, Winn-Deen E, Wolfe K, Zaveri J, Zaveri K, Abril JF, Guigo R, Campbell MJ, Sjolander KV, Karlak B, Kejariwal A, Mi H, Lazareva B, Hatton T, Narechania A, Diemer K, Muruganujan A, Guo N, Sato S, Bafna V, Istrail S, Lippert R, Schwartz R, Walenz B, Yooseph S, Allen D, Basu A, Baxendale J, Blick L, Caminha M, Carnes-Stine J, Caulk P, Chiang YH, Coyne M, Dahlke C, Deslattes Mays A, Dombroski M, Donnelly M, Ely D, Esparham S, Fosler C, Gire H, Glanowski S, Glasser K, Glodek A, Gorokhov M, Graham K, Gropman B, Harris M, Heil J, Henderson S, Hoover J, Jennings D, Jordan C, Jordan J, Kasha J, Kagan L, Kraft C, Levitsky A, Lewis M, Liu X, Lopez J, Ma D, Majoros W, McDaniel J, Murphy S, Newman M, Nguyen T, Nguyen N, Nodell M, Pan S, Peck J, Peterson M, Rowe W, Sanders R, Scott J, Simpson M, Smith T, Sprague A, Stockwell T, Turner R, Venter E, Wang M, Wen M, Wu D, Wu M, Xia A, Zandieh A, Zhu X. The sequence of the human genome. Science. 2001 Feb 16;291(5507):1304-51. doi: 10.1126/science.1058040. PMID 11181995
- [Background] Lander ES, Linton LM, Birren B, Nusbaum C, Zody MC, Baldwin J, Devon K, Dewar K, Doyle M, FitzHugh W, Funke R, Gage D, Harris K, Heaford A, Howland J, Kann L, Lehoczky J, LeVine R, McEwan P, McKernan K, Meldrim J, Mesirov JP, Miranda C, Morris W, Naylor J, Raymond C, Rosetti M, Santos R, Sheridan A, Sougnez C, Stange-Thomann Y, Stojanovic N, Subramanian A, Wyman D, Rogers J, Sulston J, Ainscough R, Beck S, Bentley D, Burton J, Clee C, Carter N, Coulson A, Deadman R, Deloukas P, Dunham A, Dunham I, Durbin R, French L, Grafham D, Gregory S, Hubbard T, Humphray S, Hunt A, Jones M, Lloyd C, McMurray A, Matthews L, Mercer S, Milne S, Mullikin JC, Mungall A, Plumb R, Ross M, Shownkeen R, Sims S, Waterston RH, Wilson RK, Hillier LW, McPherson JD, Marra MA, Mardis ER, Fulton LA, Chinwalla AT, Pepin KH, Gish WR, Chissoe SL, Wendl MC, Delehaunty KD, Miner TL, Delehaunty A, Kramer JB, Cook LL, Fulton RS, Johnson DL, Minx PJ, Clifton SW, Hawkins T, Branscomb E, Predki P, Richardson P, Wenning S, Slezak T, Doggett N, Cheng JF, Olsen A, Lucas S, Elkin C, Uberbacher E, Frazier M, Gibbs RA, Muzny DM, Scherer SE, Bouck JB, Sodergren EJ, Worley KC, Rives CM, Gorrell JH, Metzker ML, Naylor SL, Kucherlapati RS, Nelson DL, Weinstock GM, Sakaki Y, Fujiyama A, Hattori M, Yada T, Toyoda A, Itoh T, Kawagoe C, Watanabe H, Totoki Y, Taylor T, Weissenbach J, Heilig R, Saurin W, Artiguenave F, Brottier P, Bruls T, Pelletier E, Robert C, Wincker P, Smith DR, Doucette-Stamm L, Rubenfield M, Weinstock K, Lee HM, Dubois J, Rosenthal A, Platzer M, Nyakatura G, Taudien S, Rump A, Yang H, Yu J, Wang J, Huang G, Gu J, Hood L, Rowen L, Madan A, Qin S, Davis RW, Federspiel NA, Abola AP, Proctor MJ, Myers RM, Schmutz J, Dickson M, Grimwood J, Cox DR, Olson MV, Kaul R, Raymond C, Shimizu N, Kawasaki K, Minoshima S, Evans GA, Athanasiou M, Schultz R, Roe BA, Chen F, Pan H, Ramser J, Lehrach H, Reinhardt R, McCombie WR, de la Bastide M, Dedhia N, Blocker H, Hornischer K, Nordsiek G, Agarwala R, Aravind L, Bailey JA, Bateman A, Batzoglou S, Birney E, Bork P, Brown DG, Burge CB, Cerutti L, Chen HC, Church D, Clamp M, Copley RR, Doerks T, Eddy SR, Eichler EE, Furey TS, Galagan J, Gilbert JG, Harmon C, Hayashizaki Y, Haussler D, Hermjakob H, Hokamp K, Jang W, Johnson LS, Jones TA, Kasif S, Kaspryzk A, Kennedy S, Kent WJ, Kitts P, Koonin EV, Korf I, Kulp D, Lancet D, Lowe TM, McLysaght A, Mikkelsen T, Moran JV, Mulder N, Pollara VJ, Ponting CP, Schuler G, Schultz J, Slater G, Smit AF, Stupka E, Szustakowki J, Thierry-Mieg D, Thierry-Mieg J, Wagner L, Wallis J, Wheeler R, Williams A, Wolf YI, Wolfe KH, Yang SP, Yeh RF, Collins F, Guyer MS, Peterson J, Felsenfeld A, Wetterstrand KA, Patrinos A, Morgan MJ, de Jong P, Catanese JJ, Osoegawa K, Shizuya H, Choi S, Chen YJ, Szustakowki J; International Human Genome Sequencing Consortium. Initial sequencing and analysis of the human genome. Nature. 2001 Feb 15;409(6822):860-921. doi: 10.1038/35057062. PMID 11237011
- [Background] Stolerman ES, Florez JC. Genomics of type 2 diabetes mellitus: implications for the clinician. Nat Rev Endocrinol. 2009 Aug;5(8):429-36. doi: 10.1038/nrendo.2009.129. Epub 2009 Jun 30. PMID 19564886
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-N-0206.html